CLINICAL TRIAL: NCT01147172
Title: A Post Approval, Multicenter, Open-Label, Longitudinal, Uncontrolled Safety Study of Cosmetic Tissue Augmentation Product (ELEVESS™) in the Treatment of Nasolabial Folds in People of Color
Brief Title: Safety Study of Cosmetic Tissue Augmentation in People of Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anika Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTA0701
Record Dates: First submitted 2010-06-03; First posted 2010-06-22 (Estimated); Results first posted 2015-04-20 (Estimated); Last update posted 2017-10-17 (Actual); Status verified 2017-09

CONDITIONS: Wrinkles
Keywords: Nasolabial Folds; Cosmetic; Injectable Dermal Filler; Hyaluronic Acid with Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elevess (Experimental): Gel implant (dermal filler) composed of hyaluronan produced by Streptococcus equi (bacterial fermentation) that is cross-linked and suspended in phosphate buffered saline with 0.3% lidocaine HCl and 0.1% sodium metabisulfite
  Interventions: Device: Elevess

INTERVENTIONS:
Device: Elevess — Injectable gel, 0.5mL or 1.0mL material supplied in a 1.0mL pre-filled sterile glass syringe with two 30 gauge needles

SUMMARY:
Elevess is intended for all skin types. However, further study of all soft tissue fillers is needed in people of color because of the increasing use of cosmetic dermal filler products.

This study is designed to evaluate the safety of an injectable hyaluronic acid based dermal filler Elevess (Anika Therapeutics, Inc., Bedford, MA). Safety will be evaluated by incidence and severity of keloid formation and pigmentation changes, and other potential adverse events in people with Fitzpatrick skin types IV, V and VI who have elected to undergo nasolabial fold (NLF) treatment with Elevess.

1. Fitzpatrick Classification of Skin Type as: IV - Burns minimally, always tans well (moderate/light brown skin; Mediterranean, Asian, Hispanic. V - Rarely burns, tans profusely (dark brown/brown skin: Middle eastern, Latin, light skinned Black, Indian) VI - Never burns, (deeply pigmented dark brown to black skin;Black)

DETAILED DESCRIPTION:
This study is designed to be an open-label, longitudinal, uncontrolled study in a minimum of 100 subjects with Fitzpatrick scale skin type of IV, V or VI at 10 or more U.S. centers who have elected to undergo NLF treatment with intradermal (deep dermal) injection of Elevess. Subjects will be followed for a minimum of 24 weeks with visit assessments at 2, 6, 12 and 24 weeks after the last injection.

Safety: Primary Safety Endpoint assessments will be: 1) keloid formation at the site of injection at 2, 6, 12 and 24 weeks, 2) pigmentation changes at the site of injection compared to adjacent skin at 2, 6, 12 and 24 weeks, and 3) overall adverse events. A subject diary will also be collected.

Effectiveness: No formal effectiveness evaluation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick skin type of IV, V or VI.
* Bilateral nasolabial folds which, in the investigator's judgment, can be corrected with Elevess.
* Age greater or equal to 18 years.

Exclusion Criteria:

* Fitzpatrick skin type of I, II or III.
* Subject has severe allergies manifested by a history of anaphylaxis or history or presence of multiple severe allergies.
* Subject has allergies to the components of Elevess: hyaluronic acid, lidocaine, sodium metabisulfite or gram positive bacterial proteins.
* Subject has a history of severe keloids and/or hypertrophic scars.
* Subject has ever received any soft tissue augmentation in any area of the face and subject is unwilling to forgo all other soft tissue augmentation for the duration of the study.
* Subject has received any aesthetic or dermatologic treatments or procedures in any area of the face in the previous 6 months and subject is unwilling to forgo such treatments or procedures for the duration of the study.
* Subject has active facial acne lesions, severe acne scarring or pigmentation disorders at the injection site that might affect clinical assessment of the nasolabial folds.
* Subject has ever received an injection or implant of silicone in any area of the face.
* Subject has received immunosuppressive therapy, chemotherapy, or systemic corticosteroids within the last 3 months.
* Subject has a history of a connective tissue disease.
* Subject is positive for HIV/AIDS or hepatitis C.
* Subject is involved in any other research study involving an investigational product (drug, device or biologic) or a new application of an approved product, within 30 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Brandt, MD, Principal Investigator — Dermatology Research Institute, LLC; William P Coleman, MD, Principal Investigator — Private Practice; Michael Gold, MD, Principal Investigator — Tennessee Clinical Research Center; Alicia Barba, MD, Principal Investigator — International Dermatology Research, Inc.; Andrew Alexis, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center; Michael Jarratt, MD, Principal Investigator — Derm Research, Inc.; Pearl Grimes, MD, Principal Investigator — Vitiligo & Pigmentation Institute of Southern California; Marta Rendon, MD, Principal Investigator — Skin Care Research, Inc.; Eduardo Tschen, MD, Principal Investigator — Academic Dermatology Associates
Locations (9):
- United States (9):
  - Vitiligo and Pigmentation Inst of Southern California, Los Angeles, California
  - Skin Care Research, Inc., Boca Raton, Florida
  - Dermatology Research Institute, LLC, Coral Gables, Florida
  - International Dermatology Research, Miami, Florida
  - William Coleman, MD, Metairie, Louisiana
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - St Luke's Roosevelt, New York, New York
  - Tenneesee Clinical Research Center, Nashville, Tennessee
  - Derm Research, Inc., Austin, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kokelj F, Burnett JW. Treatment of a pigmented lesion induced by a Pelagia noctiluca sting. Cutis. 1990 Jul;46(1):62-4. PMID 1974491
- [Background] Linder SA, Mele JA 3rd, Harries T. Chronic hyperpigmentation from a heated mustard compress burn: a case report. J Burn Care Rehabil. 1996 Jul-Aug;17(4):351-2. doi: 10.1097/00004630-199607000-00012. PMID 8844357
- [Background] Royston SL, Wright PA, Widdowson DC, Wareham WJ, Strike PW. Adverse effects reported in epilatory ruby laser treatment. Lasers Med Sci. 2008 Jan;23(1):35-9. doi: 10.1007/s10103-007-0451-0. Epub 2007 Mar 13. PMID 17431730
- [Background] Tomita Y, Maeda K, Tagami H. Mechanisms for hyperpigmentation in postinflammatory pigmentation, urticaria pigmentosa and sunburn. Dermatologica. 1989;179 Suppl 1:49-53. doi: 10.1159/000248449. PMID 2550287

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 122 subjects were screened for the study at 9 centers. Twenty-two screen failed and 100 were were enrolled in this study. No subject who failed screening was treated during the CTA-0701 study. Of the treated subjects 96% completed the follow-up visit 24 weeks after Treatment.
Pre-assignment Details: Elevess was injected into the mid to deep dermis of each nasolabial fold. Subjects were telephoned at 72 (±24) hours to assess the subjects for possible AEs and injection site reactions. All subjects returned 14 ± 3 days after initial treatment for evaluation of AEs and to assess whether a Touch-up was needed.
Groups:
- Elevess: Gel implant (dermal filler) composed of hyaluronan produced by Streptococcus equi (bacterial fermentation) that is cross-linked and suspended in phosphate buffered saline with 0.3% lidocaine HCl and 0.1% sodium metabisulfite
  Elevess : Injectable gel, 0.5mL or 1.0mL material supplied in a 1.0mL pre-filled sterile glass syringe with two 30 gauge needles
Period: Overall Study
Arm/Group | Elevess
Started | 100
Completed | 96
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Subjects of Fitzpatrick Skin Type IV, V or VI seeking treatment of nasolabial folds with injectable hyaluronic acid gel (Elevess).
Arm/Group | Elevess
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 41
  White | 0
  More than one race | 2
  Unknown or Not Reported | 53

OUTCOME MEASURES:

1. Primary Outcome: Keloid Formation at Site of Injection
Description: Percentage of Subjects with keloid formation at the site of injection
Time Frame: 2 Weeks
Population: Safety Population
Measure: Number; unit: percentage of participants
Groups:
- Elevess: Subjects that received injection(s) of Elevess and exhibited keloid formation.
Arm/Group | Elevess
Number analyzed (Participants) | 97
percentage of participants | 0.0

2. Primary Outcome: Keloid Formation at Site of Injection
Description: Percentage of Subjects with keloid formation at the site of injection
Time Frame: 6 Weeks
Population: Safety Population
Measure: Number; unit: Percentage (%) of subjects
Arm/Group | Elevess
Number analyzed (Participants) | 97
Percentage (%) of subjects | 0.0

3. Primary Outcome: Keloid Formation at Site of Injection
Description: Percentage of Subjects with keloid formation at the site of injection
Time Frame: 12 Weeks
Population: Safety Population
Measure: Number; unit: Percentage (%) of subjects
Arm/Group | Elevess
Number analyzed (Participants) | 94
Percentage (%) of subjects | 0.0

4. Primary Outcome: Keloid Formation at Site of Injection
Description: Percentage of subjects with keloid formation at the site of injection at End of Study
Time Frame: 24 Weeks
Population: Safety Population
Measure: Number; unit: Percentage (%) of subjects
Groups:
- Elevess: Subjects that received injection(s) of Elevess and exhibited keloid formation at End of Study.
Arm/Group | Elevess
Number analyzed (Participants) | 98
Percentage (%) of subjects | 0.0

5. Primary Outcome: Pigmentation Changes at Site of Injection
Description: Percentage of Subjects with pigmentation changes at site of injection
Time Frame: 2 Weeks
Population: Safety Population
Measure: Number; unit: Percentage (%) of subjects
Groups:
- Elevess: Subjects received injection(s) and exhibited pigmentation changes at End of Study.
Arm/Group | Elevess
Number analyzed (Participants) | 97
Percentage (%) of subjects | 8.0

6. Primary Outcome: Pigmentation Changes at Site of Injection
Description: Percentage of Subjects with pigmentation changes at site of injection
Time Frame: 6 Weeks
Population: Safety Population
Measure: Number; unit: Percentage (%) of subjects
Arm/Group | Elevess
Number analyzed (Participants) | 97
Percentage (%) of subjects | 3.0

7. Primary Outcome: Pigmentation Changes at Site of Injection
Description: Percentage of Subjects with pigmentation changes at site of injection
Time Frame: 12 Weeks
Population: Safety Population
Measure: Number; unit: Percentage (%) of subjects
Arm/Group | Elevess
Number analyzed (Participants) | 94
Percentage (%) of subjects | 2.0

8. Primary Outcome: Pigmentation Changes at Site of Injection
Description: Percentage of subjects with pigmentation changes at site of injection at End of Study
Time Frame: 24 Weeks
Population: Safety Population
Measure: Number; unit: Percentage (%) of subjects
Arm/Group | Elevess
Number analyzed (Participants) | 98
Percentage (%) of subjects | 1.0

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded to 24 Weeks.
Groups:
- Safety Population: All Subjects receiving treatment of nasolabial folds (NLF) with injection of Elevess.
Arm/Group | Safety Population
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 47/100
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=100)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Eye Swelling (Eye disorders) | 1 (1)
Lip Swelling (Gastrointestinal disorders) | 1 (1)
Dental Caries (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Injection Site Discoloration (General disorders) | 10 (13)
Injection Site Dryness (General disorders) | 1 (1)
Injection Site Erythema (General disorders) | 3 (3)
Injection Site Hematoma (General disorders) | 1 (1)
Injection Site Induration (General disorders) | 5 (7)
Injection Site Irritation (General disorders) | 1 (7)
Injection Site Nodule (General disorders) | 4 (4)
Injection Site Pain (General disorders) | 4 (4)
Injection Site Pruritus (General disorders) | 1 (3)
Injection Site Scab (General disorders) | 1 (1)
Injection Site Swelling (General disorders) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Gastrointestinal Bacterial Infection (Infections and infestations) | 1 (1)
Helicobacter Pylori (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4)
Tooth Infection (Infections and infestations) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (6)
Cartilage Injury (Injury, poisoning and procedural complications) | 1 (1)
Joint Sprain (Injury, poisoning and procedural complications) | 1 (1)
Ligament Injury (Injury, poisoning and procedural complications) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bunion (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (6)
Insomnia (Psychiatric disorders) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Vasoconstriction (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less